CLINICAL TRIAL: NCT03884699
Title: Accuracy of Waferless One Stage Segmental Lefort I Maxillary Positioning in Transverse Deficiency Using CAD/CAM Patient Specific Titanium Implants (Case Series Study)
Brief Title: Waferless One Stage Segmental Lefort I Maxillary Positioning in Transverse Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Anwar Ibrahim Taman, Assistant Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3-3-7
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Lefort I Osteotomy
Keywords: Orthognathic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Segmental maxillary lefort I re-positioning (Other): Accuracy of the planned virtually re-positioned segmental Lefort I maxilla using a specifically designed patient implant, comparing the virtual plan to the actual postoperative position.
  Interventions: Procedure: Accuracy of planned transverse Maxillary distance using Mimics software after fixation using Patient specific implant

INTERVENTIONS:
Procedure: Accuracy of planned transverse Maxillary distance using Mimics software after fixation using Patient specific implant — Virtual planning: based on clinical evaluation and 3D cephalometric analysis. Virtual osteotomies mimicking segmental Lefort I and a bilateral sagittal split osteotomy.
  Designing the virtual cutting guide. Virtual movement into the desired positions of the segmented maxilla and mandible, based on: clinical evaluation, 3D cephalometric analysis and the desired occlusion.
  Once the optimal position of the maxilla is achieved, a patient specific implant will be virtually designed to fix the segmented maxilla in its new position.
  Fabrication of the cutting guide using additive manufacturing technique from polymer material.
  Fabrication of PSI from titanium alloy using additive manufacturing technique.

SUMMARY:
In Maxillary transverse deficiency, is waverless lefort I multiple pieces osteotomy using virtually planned patient specific titanium implants feasible and does it provide accuracy?

This prospective case series study evaluating the postoperative outcomes and accuracy of preoperatively planned positional changes together with virtually designed drilling and fixation guides for the waferless positioning and fixation of the multiple pieces Le Fort I of the maxilla using CAD-CAM designed patient-specific implants.

The purpose of this study is to develop and validate an orthognathic CAD/CAM patient specific implant together with template that can guide both the osteotomy and the repositioning of the maxilla during the correction of transverse maxillary deficiency.

Thus, the traditional model and the additional preparation for CAD/CAM surgical splints including scanning dental casts, and recording and moving virtual dental casts, were not required. The preoperative and laboratory procedures were simplified, and the intermediate splint technique was eliminated, so the associated potential errors were avoided.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the accuracy of planned waferless positioning of lefort I multiple piece osteotomy in maxillary deficient patients using CAD-CAM patient-specific implants together with virtually designed drilling and fixation guides.

Interventions

1. Diagnostic procedures:

   All Patients will be selected according to inclusion and exclusion criteria & Comprehensive clinical examination and understanding of patients' chief complains and needs will be carried out Preoperative patient photographs (Frontal, Profile, 45°, smile, and dental occlusion) Alginate Impressions† of upper & lower jaws for acquiring diagnostic dental casts Cone Beam Computed Topography (CBCT) for the patients §
2. Planning procedures:

Computer-aided planning: All planning will be done using specialized Mimics software** Import CBCT into virtual planning software. Segmentation: highlighting and selection of the bony anatomy based on bone density (Hounsfield Units).

3D reconstruction: virtual 3D model. CT scanning of the dental stone casts. Image fusion: to combine the virtual casts onto the 3D bony model to obtain a composite artifact-free skull model.

Virtual planning: based on clinical evaluation and 3D cephalometric analysis. Virtual osteotomies mimicking segmental Lefort I and a bilateral sagittal split osteotomy.

Designing the virtual cutting guide. Virtual movement into the desired positions of the segmented maxilla and mandible, based on: clinical evaluation, 3D cephalometric analysis and the desired occlusion.

Once the optimal position of the maxilla is achieved, a patient specific implant will be virtually designed to fix the segmented maxilla in its new position.

Fabrication of the cutting guide using additive manufacturing technique from polymer material.

Fabrication of PSI from titanium alloy using additive manufacturing technique.

3. Intra operative procedures The surgical procedures will be carried out by RT under the supervisor of AH in the Oral & Maxillofacial operating floor on the 8th floor of the faculty of Oral & Dental Medicine new building.Scrubbing and draping of the patient will be carried out in a standard fashion according to Anon 2006.

Local anesthesia (lidocaine 2%, 1/100000 adrenaline) will be injected intraorally along the incision lines for hemostasis.

Access through a vestibular intraoral incision for maxilla & Sagittal split incision for mandible will carried out. Dissection and reflection to reach the bone.

Bilateral Sagittal Split mandibular osteotomies will carried out. The osteotomy guide 2 parts will into fit the left and right side the anterior maxillary walls separately during the operation for ease of use.

Le Fort I Maxillary osteotomies will carried out using the osteotomy guide. Complete mobilization of maxillary segments. Reposition and fixation of the maxillary segments into the planned position will be done by the Patient Specific Implant (PSI) using the drilling site done by the osteotomy guide.

Reposition and fixation of the mandibular segments using bicortical screws. The incisions will be closed with continuous mattress absorbable sutures††. 4. Postoperative care & Follow up Post-operative treatment will start immediately postoperative (4 hours) Patients will start antibiotics 4 hours after the last intraoperative dose (Amoxicillin / Clavulanic acid 625 mg every 8 hours) for 5 days Patients will start analgesics (NSAIDs every 6 hours) for 3 days Mouthwash (Chlorhexidine 0.12%) will be prescribed for 2 more weeks. The patients will be scheduled for follow-up visits weekly for a month then on a monthly basis for 5 more months.

At 1 to 3 weeks postoperatively CBCT using same parameters will be ordered to calculate the difference between surgical plan and actual outcome will be evaluated.

Patient will be referred back to the orthodontist to receive his postsurgical orthodontics.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from transverse and anteroposterior maxillary discrepancy.
* Patients requiring bimaxillary orthognathic surgery.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow-up period.
* Highly motivated patients.

Exclusion Criteria:

* Patients who are younger than 14 years.
* Patients having a significant systemic disease that may affect normal healing.
* Intra-bony lesions or infections that may retard the osteotomy healing.
* Patients receiving chemo or radiotherapy.
* Known allergies or sensitivities to dental materials, including Titanium or general anesthesia agents.
* Patient with bad oral hygiene.
* Pregnant females.
* Inability to return for follow up visits.
* Refusal of participation from the patient.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Transverse dimension of maxilla on virtual plan and postoperative | 1-3 months
  8 Reference points will be chosen below the osteotomy line on the maxilla (4 dental and 4 bony), and the distances between these points and the Frankfort, the midfacial, and the coronal planes, to show the vertical, horizontal, and axial positions of the maxilla, respectively.
  These distances will be measured on the postoperative CT data and their deviations from the virtual plan will illustrate the accuracy of our procedure.
  The 4 bony reference points are :
  PF: Piriform at the widest point ; J: The junction between the maxillary tuberosity outline and the zygomatic process (63); and GPF: Greater palatine foramen.
  The 4 dental reference points are:
  A3L: Cusp of the left maxillary canine; A3R: Cusp of the right maxillary canine; A6L: Mesiobuccal cusp of the left first maxillary molar; and A6R: Mesiobuccal cusp of the right first maxillary molar.

SECONDARY OUTCOMES:
Planning & surgical times: estimated time to the actual time | 1-3 months
  Using chronometer, the time from the start of virtual plan & design, and the time of the surgery will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Taman, Msc, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No